CLINICAL TRIAL: NCT00282191
Title: Prevalence of Spasticity in Adults With Mental Retardation Residing in a Community Setting
Brief Title: Prevalence of Spasticity in Adults With Mental Retardation Living in the Community
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: David Charles, M.D., Vanderbilt University Medical Center Department of Neurology
Other Study IDs: 051220
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Mental Retardation; Spasticity
Keywords: spasticity; mental retardation
MeSH Terms: conditions — Intellectual Disability; Muscle Spasticity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This survey aims to investigate the prevalence of spasticity among adults who live in community settings in Davidson County, Tennessee. The treatment of spasticity in those who live in community homes could significantly increase a person's quality of life by allowing them to participate more independently in activities of daily living, or by making assistance easier for caregivers.

DETAILED DESCRIPTION:
The process of deinstitutionalization has transitioned a large majority of persons with developmental disabilities into the community over the past several decades, and that number will only increase going forward. There are 926 people in this region who are provided assistance through the Division of Mental Retardation Services (DMRS). People with developmental disabilities frequently have comorbidities such as spasticity that hinder their ability to participate in activities of daily living. Spasticity results from brain or spinal cord injury and can produce increased muscle tone, causing joint stiffness, contractures and pain that can interfere with recommended treatment. A previous survey conducted at Clover Bottom Developmental Center investigated care areas typically affected by spasticity, including splinting, hygiene, dressing, transfers, positioning, ambulation, and engaging in other functional activities. Pfister et al. reported the prevalence of spasticity in the developmental center to be 35% (72/205); of those people, the Survey Physician felt that 75% (54/72) would achieve a functional benefit from treatment.

Primary endpoints will assess the prevalence of spasticity in adults who reside in the community, and whether or not spasticity impacts activities of daily living. When appropriate, potential care area goals will be identified, and treatment options will be recorded. Secondary endpoints will examine whether or not participants currently receive treatment for spasticity; if so, what treatment is being used; and which care areas are most impacted by spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 and over) with mental retardation
* Living in a community home in Davidson County, Tennessee.

Exclusion Criteria:

None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with mental retardation living in community homes in Davidson County, TN.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Charles, MD, Principal Investigator — Vanderbilt University Department of Neurology
Locations (1):
- Homes, Davidson County, Tennessee, United States